CLINICAL TRIAL: NCT07356102
Title: Comparing Conventional and High-Voltage Long-Duration Pulsed Radiofrequency Applied to the Pudendal Nerve in the Treatment of Pudendal Neuralgia: A Randomized Controlled Trial
Brief Title: Conventional Versus High-Voltage Long-Duration Pulsed Radiofrequency of the Pudendal Nerve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şükriye Dadalı, Principal Investigator, Department of Pain Medicine, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-25-10056
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pudendal Neuralgia
Keywords: Pudendal Neuralgia; Pudendal Nerve; Pulsed Radiofrequency; PRF; Conventional PRF; High-Voltage Long-Duration PRF; Chronic Pelvic Pain
MeSH Terms: conditions — Pudendal Neuralgia | interventions — Drugs, Generic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. One group will receive conventional pulsed radiofrequency (PRF) of the pudendal nerve, and the other group will receive high-voltage long-duration PRF. Each participant will receive only one type of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Conventional PRF (Experimental): Conventional Pulsed Radiofrequency Description: Conventional PRF applied to the pudendal nerve at 42°C for 360 seconds, 2 Hz, 20 ms pulse width. Standard clinical procedure under sterile conditions.
  Interventions: Procedure: Intervention Type * Select the type of intervention. Procedure / Surgery Intervention Name * Enter a brief, descriptive name for the intervention. Use a non-proprietary (generic) name, if available
- Arm 2 - High-Voltage Long-Duration PRF (Experimental): High-Voltage Long-Duration Pulsed Radiofrequency Description: High-voltage, long-duration PRF applied to the pudendal nerve at 42°C for 900 seconds, voltage titrated from 40V to patient-tolerated maximum of 90V. Procedure performed under sterile conditions.
  Interventions: Procedure: High-Voltage Long-Duration Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Intervention Type * Select the type of intervention. Procedure / Surgery Intervention Name * Enter a brief, descriptive name for the intervention. Use a non-proprietary (generic) name, if available — Conventional pulsed radiofrequency (PRF) is applied to the pudendal nerve at 42°C for 360 seconds, with a pulse frequency of 2 Hz and pulse width of 20 ms. The procedure is performed under sterile conditions in the operating room with patient monitoring (blood pressure, pulse, ECG, oxygen saturation). Patients are positioned prone, the target site is sterilized, and the PRF needle is placed under fluoroscopic guidance. Bilateral symptoms are treated sequentially if present.
  Arms: Arm 1 - Conventional PRF
Procedure: High-Voltage Long-Duration Pulsed Radiofrequency — High-voltage long-duration pulsed radiofrequency (PRF) is applied to the pudendal nerve at 42°C for 900 seconds, with a pulse frequency of 2 Hz and pulse width of 20 ms. The voltage is titrated from 40V to a patient-tolerated maximum of 90V. The procedure is performed under sterile conditions in the operating room with patient monitoring (blood pressure, pulse, ECG, oxygen saturation). Patients are positioned prone, the target site is sterilized, and the PRF needle is placed under fluoroscopic guidance. Bilateral symptoms are treated sequentially if present.
  Arms: Arm 2 - High-Voltage Long-Duration PRF

SUMMARY:
This study is a single-center, prospective, randomized controlled trial evaluating two types of pulsed radiofrequency (PRF) treatment for patients with pudendal neuralgia. Pudendal neuralgia is a chronic neuropathic pain affecting the perineum and pelvic area, often causing significant discomfort and reduced quality of life.

Patients will be randomly assigned to receive either conventional PRF or high-voltage long-duration PRF applied to the pudendal nerve. The study aims to compare the clinical effectiveness, pain relief, and safety of the two treatment approaches. Participants will be monitored for pain improvement, functional outcomes, and any treatment-related side effects.

The study follows standard clinical procedures and all treatments are performed under sterile conditions with proper monitoring to ensure patient safety.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled trial aims to compare the clinical effectiveness and safety of conventional pulsed radiofrequency (PRF) versus high-voltage long-duration PRF applied to the pudendal nerve in patients with pudendal neuralgia.

Eligible patients will be randomly assigned to one of the two intervention groups. Conventional PRF will be applied at 42°C for 360 seconds, while high-voltage long-duration PRF will be applied at 42°C for up to 900 seconds, with voltage titrated from 40V to a patient-tolerated maximum of 90V. All procedures are performed under sterile conditions in an operating room with patient monitoring (blood pressure, pulse, ECG, and oxygen saturation).

Patients will be assessed for pain intensity, functional improvement, and adverse effects at scheduled follow-up visits. Bilateral symptoms will be treated sequentially if present. The study adheres to standard clinical safety procedures and no additional risk beyond routine clinical care is anticipated.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older
* Diagnosis of pudendal neuralgia according to the Nantes diagnostic criteria
* Followed at the Algology (Pain Medicine) outpatient clinic
* Chronic pudendal neuralgia refractory to conservative treatment or intolerance to conservative therapies
* Not using neuropathic pain medications, or on a stable dose for at least 3 months prior to enrollment
* Ability to comply with study procedures and follow-up visits
* Ability to understand the study information and provide written informed consent

Exclusion Criteria

* Presence of pelvic organic pathologies that may cause pudendal pain
* Pain limited only to the coccygeal, gluteal, or lower abdominal regions
* Patients with purely paroxysmal pain, isolated pruritus, or imaging findings that fully explain symptoms
* History of malignancy or autoimmune disease
* Previous surgery that may have altered the anatomy of the pudendal nerve region
* Pregnancy or suspected pregnancy
* Presence of a cardiac pacemaker or implanted electrical device
* Use of anticoagulant therapy or presence of uncorrectable coagulation disorders
* Active systemic infection or infection at the injection site
* Known hypersensitivity to metals
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Assessed by Numeric Rating Scale (NRS) | Baseline, 1 month, 3 months, and 6 months
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. The primary outcome is the change in NRS score from baseline to 6 months after treatment. Higher scores indicate greater pain intensity. NRS scores will also be recorded at 1 and 3 months to allow longitudinal comparison.

SECONDARY OUTCOMES:
Global Perceived Effect (GPE) Score | Baseline, 1 month, 3 months, and 6 months
  Patient-reported global improvement will be assessed using the Global Perceived Effect (GPE) scale, a Likert-type scale ranging from -5 to +5, where negative values indicate worsening, 0 indicates no change, and positive values indicate improvement. Higher scores indicate a better perceived outcome.
Patient Satisfaction Score | Baseline, 1 month, 3 months, and 6 months
  Patient satisfaction with treatment will be assessed using a 5-point satisfaction scale ranging from 0 (not satisfied at all) to 4 (very satisfied).
Quality of Life Assessed by Short Form-36 (SF-36) | Baseline and 6 months
  Health-related quality of life will be evaluated using the Short Form-36 (SF-36) questionnaire.
Adverse Events and Complications | From intervention to 6 months
  All procedure-related adverse events and complications will be recorded throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not shared due to institutional and legal restrictions on patient data protection.